CLINICAL TRIAL: NCT00304096
Title: Evaluation of the Safety and Immunogenicity of Vaccination With Multiple Synthetic Peptides in Participants With Advanced Breast Cancer
Brief Title: Vaccine Therapy in Treating Patients With Stage III or Stage IV Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11992; UVACC-BREAST-34; UVACC-HIT-032.7; UVACC-PRC-366-05; UVACC-GCRC-DRB001
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-02

CONDITIONS: Breast Cancer
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; male breast cancer; invasive lobular breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Carcinoma, Lobular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1: Receiving Hormone Therapy (Experimental): Patients treated with 9 peptide vaccine who received hormone therapy
  Interventions: Biological: synthetic breast cancer peptides-tetanus toxoid-Montanide ISA-51 vaccine
- Stratum 2: Not receiving hormone therapy (Experimental): Patients receiving 9 peptide vaccine who did not receive hormone therapy
  Interventions: Biological: synthetic breast cancer peptides-tetanus toxoid-Montanide ISA-51 vaccine

INTERVENTIONS:
Biological: synthetic breast cancer peptides-tetanus toxoid-Montanide ISA-51 vaccine

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Giving booster vaccinations may make a stronger immune response and kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy in treating patients with stage III or stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety of a vaccine comprising multiple synthetic breast cancer-associated peptides and a tetanus toxoid helper peptide emulsified in Montanide ISA-51 in patients with stage III or IV adenocarcinoma of the breast.
* Determine, preliminarily, the frequency of immune responses against the 9 class I MHC-restricted peptides in patients treated with the vaccine.
* Determine, preliminarily, the cytotoxic responses of T-cells to allogeneic breast cancer cells and autologous breast cancer cells (when available).

OUTLINE: This is an open-label study.

Patients receive peptide vaccine comprising 9 synthetic breast cancer peptides and tetanus toxoid helper peptide emulsified in Montanide ISA-51 subcutaneously and intradermally once daily on days 1, 8, 15, 36, 57, and 78 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed adenocarcinoma of the breast

  * Stage III or IV disease
  * Primary or recurrent disease
  * Invasive lobular carcinoma allowed
* HLA-A1, -A2, -A3, or -A31 positive
* Underwent and recovered from prior primary therapy

  * Patients with no clinical or radiological evidence of disease who had a previous diagnosis of stage III or IV breast cancer must have undergone prior antineoplastic therapy including, but not limited to, surgery, chemotherapy, and radiotherapy within the past 36 months
* Must have at least one undissected axillary and/or inguinal lymph node basin
* No history of brain metastases
* Hormone receptor status

  * Estrogen receptor-positive or -negative tumor

PATIENT CHARACTERISTICS:

* ECOG performance status of 0 or 1
* Body weight > 110 lbs (without clothes)
* Male or female
* Menopausal status not specified
* Absolute neutrophil count > 1000/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL
* Hemoglobin A1c < 7%
* AST and ALT ≤ 2.5 x upper limit of normal (ULN)
* Bilirubin ≤ 2.5 x ULN
* Alkaline phosphatase ≤ 2.5 x ULN
* Creatinine ≤ 1.5 x ULN
* HIV negative
* Hepatitis C negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known or suspected allergies to any component of the vaccine
* No active infection requiring antibiotics
* No New York Heart Association class III or IV heart disease
* No autoimmune disorders requiring cytotoxic or immunosuppressive therapy or autoimmune disorders with visceral involvement, except the following:

  * Laboratory evidence of autoimmune disease (e.g., positive ANA titer) without symptoms
  * Clinical evidence of vitiligo
  * Other forms of depigmenting illness
  * Mild arthritis requiring nonsteroidal antiinflammatory drugs
* No medical contraindication or potential problem that would preclude study participation

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior surgery
* More than 4 weeks since prior and no concurrent chemotherapy and radiotherapy
* More than 4 weeks since prior and no concurrent allergy desensitization injections
* More than 4 weeks since prior parenteral, oral, or inhaled corticosteroids

  * No concurrent inhaled steroids (e.g., Advair® or triamcinolone acetonide)
  * Prior or concurrent topical corticosteroids allowed
* More than 4 weeks since prior and no concurrent growth factors (e.g., epoetin alfa, darbepoetin alfa, or pegfilgrastim)
* More than 4 weeks since prior and no concurrent other investigational medication
* More than 4 weeks since prior and no concurrent other agents with putative immunomodulating activity except for non-steroidal anti-inflammatory agents
* Prior and concurrent hormonal therapy (e.g., tamoxifen, raloxifene, toremifene, fulvestrant, letrozole, anastrozole, or exemestane) allowed
* No prior vaccination with any synthetic peptides in this protocol

  * Vaccines for infectious disease (e.g., influenza) allowed, provided they are administered ≥ 2 weeks prior to or ≥ 2 weeks after study vaccine
* Short term therapy for acute conditions not related to breast cancer allowed
* No concurrent illegal drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-12; Primary Completion 2007-06 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Brenin, MD, FACS, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University of Virginia Dec 13, 2005 to May 6, 2008
Pre-assignment Details: 12 participants were registered to the study and 11 received vaccines. One participant was not compliant and did not receive vaccine.
Groups:
- Stratum 1: Received Hormonal Therapy: Participants received hormonal therapy
- Stratum 2: Had Not Received Hormonal Therapy: Participants had not received hormonal therapy
Period: Overall Study
Arm/Group | Stratum 1: Received Hormonal Therapy | Stratum 2: Had Not Received Hormonal Therapy
Started | 6 | 5
Completed | 6 | 5 (6 patients enrolled, 1 not treated)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1: Received Hormonal Therapy | Stratum 2: Had Not Received Hormonal Therapy | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 2 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 56.7 (5.75) | 59.6 (14.47) | 58.0 (10.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experienced Dose-limiting Adverse Events
Description: Safety of the 9-peptide mixture if fewer than 33% of patients experience a dose-limiting toxicity
Time Frame: 30 days post administration of last vaccine
Measure: Number; unit: participants
Arm/Group | Stratum 1: Received Hormonal Therapy | Stratum 2: Had Not Received Hormonal Therapy
Number analyzed (Participants) | 6 | 5
participants | 1 | 0

2. Secondary Outcome: The Number of Participants With T-cell Responses Against the Vaccine as Measured by Elispot Assay After 14 Day in Vitro Sensitization
Time Frame: Days 1-78
Measure: Number; unit: participants
Arm/Group | Stratum 1: Received Hormonal Therapy | Stratum 2: Had Not Received Hormonal Therapy
Number analyzed (Participants) | 6 | 5
participants | 5 | 3

ADVERSE EVENTS:
Time Frame: 30 days post last vaccine
Arm/Group | Stratum 1: Received Hormonal Therapy | Stratum 2: Had Not Received Hormonal Therapy
Serious Adverse Events (participants affected / at risk) | 1/6 | 0/5
Other Adverse Events (participants affected / at risk) | 1/6 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1: Received Hormonal Therapy (N=6) | Stratum 2: Had Not Received Hormonal Therapy (N=5)
Fever (General disorders) | 1 (1) | 0 (0) — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1: Received Hormonal Therapy (N=6) | Stratum 2: Had Not Received Hormonal Therapy (N=5)
Fatigue (General disorders) | 1 (1) | 0 (0) — Grade 3 fatigue was an expected event.
Pain, headache (General disorders) | 0 (0) | 1 (1) — Grade 3 headache was an expected event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes